CLINICAL TRIAL: NCT01272583
Title: Effects of 6 Weeks Treatment With a Dipeptidyl Peptidase 4 Inhibitor on Counterregulatory and Incretin Hormones During Acute Hypoglycaemia in Patients With Type 1 Diabetes: a Randomized Double Blind Placebo-controlled Cross-over Study
Brief Title: Dipeptidyl Peptidase-4 Inhibitors and Alpha-cell Recovery
Acronym: DARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, F Holleman, PhD, MD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: DARE_2010
Record Dates: First submitted 2011-01-05; First posted 2011-01-10 (Estimated); Results first posted 2014-02-17 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-02

CONDITIONS: Type 1 Diabetes; Hypoglycemia
Keywords: Type 1 diabetes; DPP-4 inhibitor; Glucagon
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence A (sitagliptin→placebo) (Other): Cross-over, both arms reveived the same intervention in different order.
  Interventions: Drug: Sitagliptin; Drug: Placebo
- Sequence B (placebo→sitagliptin) (Other): Cross-over, both arms reveived the same intervention in different order.
  Interventions: Drug: Sitagliptin; Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin — 100 mg once daily for six weeks
  Other Names: Januvia
Drug: Placebo — placebo, once daily for six weeks

SUMMARY:
Hypoglycaemia is a well-known complication of insulin treated diabetes. The counterregulatory response to hypoglycaemia, with glucagon as the most important mediator, is initially diminished within a few years of onset of Type 1 diabetes and subsequently lost and thus increasing the risk of hypoglycaemia. Dipeptidyl Peptidase (DPP)-4 inhibitors augment the glucagon response to insulin-induced hypoglycaemia in type 2 diabetes. The investigators hypothesize that treatment with a DPP-4 inhibitor in patients with type 1 diabetes will recover the alpha cell response to hypoglycaemia.

DETAILED DESCRIPTION:
The 16 type 1 patients will be randomised to one of two treatment sequences: DPP-4 inhibitor followed by placebo or placebo followed by a DPP-4 inhibitor. Each treatment period lasts 6 weeks, so all patients will receive treatment for 12 weeks in total. Induction of hypoglycaemia will take place at 0 weeks, 6 weeks and 12 weeks to determine the glucagon response.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes Mellitus 5-20 years duration
* C-peptide negative
* Willing and able to give written informed consent

Exclusion Criteria:

* Impaired awareness of hypoglycaemia
* BMI > 27 kg/m2
* Evidence of severe diabetes complications (autonomic neuropathy, macroalbuminuria, proliferative retinopathy)
* Acute illness within 3 months before the study
* Significant renal impairment (creatinine clearance < 50ml/min)
* Use of beta-adrenoreceptor blockers
* Cardiac history (previous arrhythmia)
* History of epilepsy

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frits Holleman, MD,PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants came to the Academic Medical Center in Amsterdam for a screening visit to determine eligibility for the study.
Pre-assignment Details: Patients were excluded if they were found to have impaired awareness of hypoglycaemia, had a history of seizures, cardiac arrhythmia (or used beta-adrenoreceptor blockers) and/or acute infection in the 12 weeks before the study, or evidence of severe diabetes complications (autonomic neuropathy, nephropathy or proliferative retinopathy).
Groups:
- Sequence A (Sitagliptin→Placebo); Sequence B (Placebo→Sitagliptin): Cross-over, both arms reveived the same intervention in different order.
  Sitagliptin : 100 mg once daily for six weeks
  Placebo : placebo, once daily for six weeks
Period: Overall Study
Arm/Group | Sequence A (Sitagliptin→Placebo) | Sequence B (Placebo→Sitagliptin)
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence A (Sitagliptin→Placebo) | Sequence B (Placebo→Sitagliptin) | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30.5 (26.3-39) [26.3 to 39] | 33.5 (27.8-40.8) [27.8 to 40.8] | 31.5 (27.0-40.0) [27.0 to 40.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  Netherlands | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Glucagon Response to Acute Hypoglycaemia
Description: Change in glucagon concentration from the initialisation phase to 40 minutes after occurrence of the autonomic reaction to hypoglycaemia
Time Frame: Change from initialisation phase to 40 minutes after onset of hypoglycaemia
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | Baseline | Sitagliptin Treatment | Placebo
Number analyzed (Participants) | 16 | 16 | 16
pmol/L | 1.33 [-0.67 to 2.67] | 1.0 [-0.67 to 2.67] | 1.33 [-1.00 to 2.33]
Statistical Analysis 1: Comparison: Baseline vs Sitagliptin Treatment vs Placebo; Test type: Superiority or Other; p = 1.0, ANOVA; The Friedman Test was used for ANOVA

2. Secondary Outcome: Intact and Total Glucagon Like Peptide-1 (GLP-1), Intact and Total Gastric Inhibitory Peptide (GIP) Response to Acute Hypoglycaemia
Description: Area under the curve (AUC) from onset of the autonomic response to hypoglycaemia to 40 minutes after onset of the autonomic response. AUC values were calculated by the trapezoid method.
Time Frame: 0, 10, 20, 40 minutes
Measure: Median (Inter-Quartile Range); unit: pmol*minutes/L
Arm/Group | Baseline | Sitagliptin Treatment | Placebo
Number analyzed (Participants) | 16 | 16 | 16
pmol*minutes/L
  GLP-1 intact | 2.000 [0.0000 to 15.50] | 43.50 [12.00 to 81.50] | 4.500 [0.0000 to 21.00]
  GLP-1 total | 562.2 [435.0 to 623.8] | 555.0 [450.0 to 611.3] | 552.5 [433.8 to 596.3]
  GIP intact | 455.0 [361.3 to 513.8] | 490.0 [461.3 to 630.0] | 452.5 [435.0 to 532.5]
  GIP total | 302.5 [201.3 to 436.3] | 285.0 [160.0 to 367.5] | 342.5 [238.8 to 497.5]
Statistical Analysis 1: Comparison: Baseline vs Sitagliptin Treatment vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA — GLP-1 intact; The Friedman Test was used for ANOVA
Statistical Analysis 2: Comparison: Baseline vs Sitagliptin Treatment vs Placebo; Test type: Superiority or Other; p = 0.98, ANOVA — GLP-1 Total; The Friedman Test was used for ANOVA
Statistical Analysis 3: Comparison: Baseline vs Sitagliptin Treatment vs Placebo; Test type: Superiority or Other; p = 0.049, ANOVA — GIP intact; The Friedman Test was used for ANOVA
Statistical Analysis 4: Comparison: Baseline vs Sitagliptin Treatment vs Placebo; Test type: Superiority or Other; p = 0.44, ANOVA — GIP total; The Friedman Test was used for ANOVA

3. Secondary Outcome: Epinephrine Response to Acute Hypoglycaemia
Description: as for outcome 2
Time Frame: 0, 10, 20, 40 minutes
Measure: Median (Inter-Quartile Range); unit: nmol*minutes/L
Arm/Group | Baseline | Sitagliptin Treatment | Placebo
Number analyzed (Participants) | 16 | 16 | 16
nmol*minutes/L | 36.1 [31.1 to 62.5] | 32.6 [17.0 to 65.0] | 58.7 [34.8 to 71.3]
Statistical Analysis 1: Comparison: Baseline vs Sitagliptin Treatment vs Placebo; Test type: Superiority or Other; p = 0.14, ANOVA; The Friedman Test was used for ANOVA

4. Primary Outcome: Glucagon Response to Acute Hypoglycaemia
Description: as for outcome 2
Time Frame: 0, 10, 20 and 40 minutes
Measure: Median (Inter-Quartile Range); unit: pmol*minutes/L
Arm/Group | Baseline | Sitagliptin Treatment | Placebo
Number analyzed (Participants) | 16 | 16 | 16
pmol*minutes/L | 120 [90 to 215] | 125 [20 to 215] | 120 [85 to 200]
Statistical Analysis 1: Comparison: Baseline vs Sitagliptin Treatment vs Placebo; Test type: Superiority or Other; p = 0.98, ANOVA; The Friedman Test was used for ANOVA

5. Secondary Outcome: Norepinephrine Response to Acute Hypoglycaemia
Description: as for outcome 2
Time Frame: 0, 10, 20, 40 minutes
Measure: Median (Inter-Quartile Range); unit: nmol*minutes/L
Arm/Group | Baseline | Sitagliptin Treatment | Placebo
Number analyzed (Participants) | 16 | 16 | 16
nmol*minutes/L | 70.0 [52.5 to 88.1] | 62.5 [44.9 to 73.0] | 62.3 [49.1 to 72.5]
Statistical Analysis 1: Comparison: Baseline vs Sitagliptin Treatment vs Placebo; Test type: Superiority or Other; p = 0.22, ANOVA; The Friedman Test was used for ANOVA

6. Secondary Outcome: Growth Hormone Response to Acute Hypoglycaemia
Description: as for outcome 2
Time Frame: 0, 10, 20, 40 minutes
Measure: Median (Inter-Quartile Range); unit: mU*minutes/L
Arm/Group | Baseline | Sitagliptin Treatment | Placebo
Number analyzed (Participants) | 16 | 16 | 16
mU*minutes/L | 1299 [313.5 to 2560] | 261.5 [47 to 1499] | 1406 [781 to 2626]
Statistical Analysis 1: Comparison: Baseline vs Sitagliptin Treatment vs Placebo; Test type: Superiority or Other; p = 0.01, ANOVA; The Friedman Test was used for ANOVA
Statistical Analysis 2: Comparison: Sitagliptin Treatment vs Placebo; Test type: Superiority or Other; p < 0.05, Dunn's Multiple Comparison Test; Post Hoc testing

7. Secondary Outcome: Cortisol Response to Acute Hypoglycaemia
Description: as for outcome 2
Time Frame: 0, 10, 20, 40 minutes
Measure: Median (Inter-Quartile Range); unit: mU*minutes/L
Arm/Group | Baseline | Sitagliptin Treatment | Placebo
Number analyzed (Participants) | 16 | 16 | 16
mU*minutes/L | 14480 [11300 to 17180] | 13190 [10920 to 18680] | 14800 [8985 to 19160]
Statistical Analysis 1: Comparison: Baseline vs Sitagliptin Treatment vs Placebo; Test type: Superiority or Other; p = 0.76, ANOVA; The Friedman Test was used for ANOVA

8. Secondary Outcome: Symptomatic Hormone Responses to Acute Hypoglycaemia.
Description: The symptomatic responses to hypoglycaemia were assessed using a standard validated symptom questionnaire adapted for experimental hypoglycaemia (McCrimmon et al (2003) Diabet.Med. 20: 507-509). A 7-point Likert scale (1=symptom absent; 7=symptom experienced with great intensity) was used to score presence and intensity of autonomic and neuroglycopenic symptoms of hypoglycaemia. Symptom scores were obtained during the initialisation phase, at occurrence of autonomic reaction and again 30 minutes later. For analyses the scale was considered as a continuous variable.
Time Frame: Change from baseline symptomatic response at hypoglycaemia and 30 minutes after hypoglycaemia
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Baseline | Sitagliptin Treatment | Placebo
Number analyzed (Participants) | 16 | 16 | 16
units on a scale
  Autonomic symptoms score | 1.7 [1.7 to 2.9] | 1.3 [1.0 to 2.6] | 1.5 [1.0 to 2.2]
  Neurologic symptoms score | 2.1 [1.7 to 3.4] | 2.4 [1.7 to 3.8] | 2.1 [1.5 to 3.3]

ADVERSE EVENTS:
Arm/Group | Baseline | Sitagliptin Treatment | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less